CLINICAL TRIAL: NCT06123234
Title: Randomised Double-blind Active vs. Placebo Clinical Trial on the Effect of the Food Effect of the Food Supplement Enterokind® Junior on Irritable Bowel Syndrome (IBS) in Children
Brief Title: Randomised Double-blind Active vs. Placebo Clinical Trial on the Effect of a Food Supplement on IBS in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENTJR
Record Dates: First submitted 2023-06-19; First posted 2023-11-08 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: Randomized double blind verum vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: different batch code assigned to products, same labeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Partecipants received a food supplement with probiotics, chamomile, vitamin A, vitamin D in single-dose vials every day for 60 days.
  Interventions: Dietary Supplement: Verum
- Placebo (Placebo Comparator): Placebo does not contain any active ingredients. Partecipants received placebo in single-dose vials every day for 60 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Verum — Food supplement in single-dose vials
  Arms: Verum
Other: Placebo — Food supplement in single-dose vials
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test a food supplement in children of 3-17 years with IBS. The main questions it aims to answer are:

* Is the tested supplement able to improve and/or reduce IBS-related symptoms?
* After administration of the food supplement, how does the state of intestinal inflammation improve?
* Is the gut microbiota modified?

Participants will take the food supplement every day for 2 months. After 30 days and after 60 days, they will be visited from the gastroenterologist.

* They have to fill in the questionnaire and the symptom's diary weekly and deliver it to the gastroenterologist during the visits
* At the first visit, they will collect the faecal sample for the analysis of inflammatory markers and gut microbiota
* After 30 days, they will collect the faecal sample for the analysis of inflammatory markers
* After 60 days, they will collect the faecal sample for the analysis of gut microbiota Researchers will compare with placebo to see if the product is effective.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a functional gastrointestinal disorder characterised essentially by abdominal pain and alterations in bowel movements. IBS is linked to a sensory and intestinal motor dysfunction, to the genesis, clinical presentation and evolution of which both medical factors (e.g. infection, inflammation, trauma, etc.) and psychosocial factors (stress, anxiety, depression, abuse, etc.) contribute. In recent decades, the prevalence of IBS, which is common in adults, has also increased in paediatric patients with rates ranging from 7 to 21%.

Due to the persistence, recurrence and intensity of pain and bowel disorders, IBS has a significant impact on patients' daily activities and quality of life. Due to the multifactorial nature of the disorder, the treatment of IBS is not simple. Supplementation with probiotic bacteria can help restore the correct state of intestinal eubiosis by repopulating the microbiota with those bacterial species that are deficient in IBS sufferers.

The formula of the product to be tested in this study contains L. acidophilus and L. reuteri and is supplemented with a dry extract of chamomile titrated in apigenin, vitamin A and vitamin D3. The product under study, therefore, is specially formulated with active ingredients and components that, based on the available literature and scientific data, can reasonably be expected to help improve intestinal inflammatory conditions and play a therapeutic role in IBS.

The aim of the study is to evaluate the effect of the dietary supplement on IBS diagnosed according to Rome IV criteria in children in the age group 3-17 years. The main objective (primary end-point) will be to evaluate the short (30 days) and medium (60 days) term effects of the product. For this purpose, a scoring questionnaire (SGARC-Subject's Global Assessment of Relief for Children) will be administered to assess relief with respect to these symptoms. All subjects who have a decrease of at least 1 point in their questionnaire score compared to the beginning of the study will be considered as "Responders". Taking into account a probable 40% Responder in the control group due to the placebo effect, the expected benefit in the active group is an improvement, compared to the initial condition, in at least 70% of the subjects (30% more Responder than placebo). As a secondary end-point, the reduction of the most common symptoms related to IBS (abdominal pain and bloating, stool characteristics, etc.) will also be assessed by means of a scoring questionnaire. Further secondary end-points will be the evaluation of the influence of the product on both the inflammatory state and the intestinal microbial populations (microbiota).

Patients will be divided into 2 groups of 50 subjects each, who will be given alternately, according to a randomisation list, the study product containing probiotics, chamomile extract and vitamins A and D3, and a placebo product, containing excipients, for 60 days. The study involves an initial visit with the referring doctor during which recruitment will take place, followed by two further visits, one after 30 and one after 60 days of taking the product.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting symptoms of IBS according to Rome IV criteria.
* Presence of functional disorders according to assessment questionnaire with a score of 2 or more.
* Age between 3 and 17 years and 11 months.
* Willingness of the subject/parent to participate in the study.
* Willingness of the subject/parent to complete the questionnaire.
* Willingness of subject/parent to use only the product to be tested during the duration of the study.
* Willingness of the subject/parent not to use similar products during the duration of the study.
* Parent's signature of informed consent.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria.
* Subjects considered unfit by the referring physician.
* Subjects with suspected or confirmed sensitivity to one or more components of the product.
* Subjects with psychiatric comorbidities.
* Subjects with serious illnesses.
* Subjects with differential diagnoses (functional dyspepsia, coeliac disease, IBD, food intolerances, individual hypersensitivities).
* Subjects undergoing ongoing pharmacological treatment, inherent to the disease (e.g. spasmolytics etc.).
* Subjects who have recently (two weeks or less) undergone antibiotic therapy
* Subjects with other concomitant diseases (immune, infectious, respiratory or gastro-intestinal).
* Subjects with growth restriction.
* Subjects with congenital malformations.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the relief of IBS related symptoms | T0 (first visit - day 0), T30 days, T60 days
  Evaluation of the relief of IBS related symptoms by means of a questionnaire to be completed during visits, which follows SGARC (Subject's Global Assessment Relief for Children) validated 5-points scale (from 0 to 4, where 0 = complete relief and 4 = worsening).
Evaluation of the reduction of IBS related symptoms | T0 (first visit - day 0), T30 days, T60 days
  Evaluation of the reduction of IBS related symptoms by means of a 2-questions questionnaire to be completed during visits

SECONDARY OUTCOMES:
Variation of inflammatory markers and of the gut microbiota | T0 (first visit - day 0), T30 days
  variation of faecal inflammatory markers calprotectin, TNFα and zonulin; effect of the product on modulation of the gut microbiota assessed by metagenomics analysis.
Metagenomic analysis of the gut microbiota | T0 (first visit - day 0), T 60 days
  Metagenomic analysis of the gut microbiota: DNA extraction, amplification and sequencing of 16S r-DNA and subsequent analysis by Next Generation Sequencing (NGS)

CONTACTS AND LOCATIONS:
Locations (1):
- Gioacchino Calapai, Messina, Italy